CLINICAL TRIAL: NCT01804036
Title: A Pilot Study of Two Contrasting Intervention Programs for Sleep Management
Brief Title: Two Contrasting Interventions for Sleep Management
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Evans Army Community Hospital (Other)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBNet-193532-1
Record Dates: First submitted 2013-02-28; First posted 2013-03-05 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Primary Insomnia; Secondary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem (Ambien) Treatment (Active Comparator): A three week treatment of Zolpidem
  Interventions: Drug: Zolpidem
- Mind-Body Bridging (Experimental): An awareness training program using mindfulness-based techniques.
  Interventions: Behavioral: Mind-Body Bridging

INTERVENTIONS:
Drug: Zolpidem — Week 1: 10 mg Zolpidem daily for 1 week, Week 2: 10 mg Zolpidem daily for one week, taken as needed, Week 3: 5 mg Zolpidem daily for 1 week, taken as needed.
  Other Names: Ambien
  Arms: Zolpidem (Ambien) Treatment
Behavioral: Mind-Body Bridging — An awareness training program. One 2 hr class per week for 3 weeks - 2 hours per session
  Other Names: Awareness Training
  Arms: Mind-Body Bridging

SUMMARY:
This study will determine whether Mind-Body Bridging (MBB), a mindfulness training program is more effective than a common sleep medication, Zolpidem, in treating insomnia. It will also investigate whether MBB is additionally beneficial for co-morbid conditions such as stress, PTSD, depression, etc, compared with that of Zolpidem.

DETAILED DESCRIPTION:
Sleep disturbance in active duty military personnel is highly prevalent and contributes to reduced performance of military duties. Under extreme conditions, army personnel could endanger themselves and their comrades. Increasingly, non-pharmacological treatments for insomnia are showing promise as complementary and alternative medicine treatments. Many of these awareness training programs (ATPs) perform as well as, or even better than, medications. This study will determine whether Mind-Body Bridging (MBB), an ATP that teaches awareness/mindfulness and cognitive skills, is more effective than a common sleep medication, Zolpidem. The study will also determine whether MBB exhibits additional benefits in co-morbid mental health conditions, including, stress, PTSD, depression, etc, compared with that of Zolpidem. This will offer soldiers additional treatment options for insomnia in the hope that it will improve both sleep and other common comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* primary insomnia
* secondary insomnia
* requiring sleep medication (Zolpidem) for a three-week trial.
* active duty military service member stationed at Fort Carson.

Exclusion Criteria:

* secondary insomnia to a likely medical condition, such as sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, and other sleep disorders, which are not appropriately treatable with sleep medication.
* treated for sleep problems using sleep medications which include Lunesta, Ambien, Ambien Controlled Release (CR), Seroquel, Trazodone or Remeron
* major psychopathology (i.e., schizophrenia)
* severe depression within the past 90 days
* suicidal ideation within the past 90 days
* psychiatrically hospitalized within the past 90 days
* uncontrolled hypertension or diabetes
* pregnancy
* previous use of Zolpidem proved to be ineffective or to cause other unwanted side effects
* actively abusing controlled substances
* enrolled in another study

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2013-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Evans Army Community Hospital, Colorado Springs, Colorado
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Mind-Body Bridging, 41 participants consented, but one participant did not provide baseline assessment data; consequently, 40 Mind-Body Bridging participants' baseline data were included in the analyses.
Groups:
- Zolpidem (Ambien) Treatment: A three week treatment of Zolpidem
  Zolpidem:
  Week 1: half dose of Zolpidem on the first night (5 mg: males/2.5 mg: females), remaining six nights, 5-10 mg (males), 2.5-5 mg (females) nightly Week 2: half or full dose, as needed. Week 3: requested to taper off sleep medication with half-dose, as needed.
Period: Overall Study
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Started | 31 | 41
Completed | 18 | 21
Not Completed | 13 | 20

BASELINE CHARACTERISTICS:
Population: In Mind-Body Bridging, 41 participants consented, but one participant did not provide baseline assessment data; consequently, 40 Mind-Body Bridging participants' baseline data were included in the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging | Total
Number analyzed (Participants) | 31 | 40 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (8.2) | 30.1 (6.9) | 30.0 (7.4)
Sex/Gender, Customized [Number; unit: participants]
  Males | 5 | 5 | 10
  Females | 25 | 35 | 60
  Not Provided | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Measures of Sleep Using Medical Outcomes Study -Sleep Scale, From Baseline at 1-week Follow-up
Description: Medical Outcomes Study - sleep scale. A 12-item validated questionnaire evaluating sleep outcomes over the past 7 days. The subscale Sleep Problems Index - II, is reported, range is 0-100. The greater the value the worse the sleep problems. In the present study, the greater the change from baseline the greater the improvement in sleep problems.
Time Frame: Baseline, 1-week follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 15.8 [9.1 to 22.4] | 16.1 [9.3 to 22.8]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.84, ANCOVA

2. Primary Outcome: Change in Subjective Measures of Sleep Using Medical Outcomes Study -Sleep Scale, From Baseline at 2 Month Follow-up
Description: as for outcome 1
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 29.38 [22.0 to 36.75] | 21.04 [13.97 to 28.11]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.11, ANCOVA

3. Primary Outcome: Change in Insomnia Severity Index, From Baseline at 1-week Follow-up
Description: Insomnia Severity Index - A 7-item validated questionnaire evaluating severity of insomnia symptoms over the past 7 days. The total score is reported with a range of 0-28. The greater the value the greater the insomnia severity. In the present study, the greater the change from baseline the greater the improvement in insomnia severity.
Time Frame: Baseline, 1-week follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 4.3 [2.2 to 6.3] | 4.0 [2.0 to 5.9]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.95, ANCOVA

4. Primary Outcome: Change in Insomnia Severity Index, From Baseline at 2 Month Follow-up
Description: as for outcome 3
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 9.34 [7.0 to 11.72] | 6.38 [4.11 to 8.66]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.08, ANCOVA

5. Primary Outcome: Change in Total Sleep Time Using a Sleep Diary, From Baseline at 1-week Follow-up
Description: Sleep Diary - 7 days of data collection. Total Sleep Time (TST, in min.): The amount of time asleep, calculated from the time of falling asleep to waking up. Range 0 - 24 hr. The greater the value the more total sleep was obtained.
Time Frame: Baseline, 1-week follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | 69.6 [36.0 to 103.1] | 38.3 [4.8 to 71.9]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.20, ANCOVA

6. Primary Outcome: Change in Total Sleep Time Using a Sleep Diary, From Baseline at 2 Month Follow-up
Description: Sleep Diary - 7 days of data collection; Total Sleep Time (TST, in min.): The amount of time asleep, calculated from the time of falling asleep to waking up. Range 0 - 24 hr. The greater the value the more total sleep was obtained.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | 74.14 [33.8 to 114.5] | 29.9 [-10.4 to 70.1]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.13, ANCOVA

7. Primary Outcome: Change in Sleep Onset Latency Using a Sleep Diary, From Baseline at 1-week Follow-up
Description: Sleep Diary - 7 days of data collection; Sleep Onset Latency (SOL, in min.): The time to fall asleep, calculated from the time of turning out the light to falling asleep. Range 0 - 24 hr. A negative value reflects an improvement in SOL at the 1-week follow-up.
Time Frame: Baseline, 1-week follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | -5.9 [-17.2 to 5.4] | -11.1 [-22.6 to 0.4]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.52, ANCOVA

8. Primary Outcome: Change in Sleep Onset Latency Using a Sleep Diary, From Baseline at 2 Month Follow-up
Description: Sleep Diary - 7 days of data collection; Sleep Onset Latency (SOL, in min.): The time to fall asleep, calculated from the time of turning out the light to falling asleep. Range 0 - 24 hr. A negative value reflects an improvement in SOL at the 2-month follow-up.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | -7.5 [-21.4 to 6.3] | -13.7 [-27.6 to 0.2]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.54, ANCOVA

9. Primary Outcome: Change in Waking After Sleep Onset Using a Sleep Diary, From Baseline at 1-week Follow-up
Description: Sleep Diary - 7 days of data collection; Waking After Sleep Onset (WASO, in min.): The duration of awakenings throughout the night, calculated after falling asleep to before the last awakening of waking up and not going back to sleep. Range 0 - 24 hr. A negative value reflects improvement in WASO at the 1-week follow-up.
Time Frame: Baseline, 1-week follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | -4.3 [-8.8 to 0.2] | -4.0 [-8.5 to 0.5]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.94, ANCOVA

10. Primary Outcome: Change in Waking After Sleep Onset Using a Sleep Diary, From Baseline at 2 Month Follow-up
Description: Sleep Diary - 7 days of data collection; Waking After Sleep Onset (WASO, in min.): The duration of awakenings throughout the night, calculated after falling asleep to before the last awakening of waking up and not going back to sleep. Range 0 - 24 hr. A negative value reflects improvement in WASO at the 2-month follow-up.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
minutes | -4.8 [-10.4 to 0.9] | -4.5 [-10.2 to 1.2]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.95, ANCOVA

11. Secondary Outcome: PTSD Check List (PCL) - Military (PCL-M)
Description: The PCL-M is a well-validated 17-item self-report measure to assess PTSD severity among military personnel; both male and female, to assess military-related PTSD. Reliability evidence is very good. Items are based on DSM criteria (DSM-IV criteria for this version) and are rated on a 5-point Likert-type scale that allows the derivation of a quantifiable total score.Range is 0-85, the greater the value the worse the PTSD reported symptoms.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 35.9 [31.5 to 40.3] | 38.0 [34.1 to 41.8]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.49, ANCOVA

12. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D is one of the most commonly validated screening tests for helping an individual to determine his or her depression quotient. The 20-item test measures depressive feelings and behaviors during the past week. Each item is summed to obtain a CES-D total score ranging from 0 to 60; higher scores indicate more severe depressive symptoms. A total score of 16 or higher was identified in early studies as indicative of individuals with depressive illness.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 19.5 [16.8 to 22.1] | 24.5 [22.2 to 26.9]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p < 0.01, ANCOVA

13. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: One of the few well-validated measures of resilience is the Connor-Davidson Resilience Scale (CD-RISC), comprising 25 items. All items are summed to obtain a CD-RISC total score ranging from 0-100, with greater total scores indicating greater resilience.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 72.9 [68.0 to 77.7] | 62.3 [58.0 to 66.6]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p < 0.01, ANCOVA

14. Secondary Outcome: Mindfulness Assessment (Five-facet Mindfulness Questionnaire; FFMQ)
Description: This is a validated questionnaire which tracks how facets of mindfulness may develop over time. It has 39 items and divides into 5 factors representing the various aspects of mindfulness. The range is 0-195. The greater the value the greater an individual's mindfulness level.
Time Frame: Baseline, 2 month follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Number analyzed (Participants) | 31 | 40
units on a scale | 126.9 [120.0 to 133.8] | 120.1 [114.3 to 125.8]
Statistical Analysis 1: Comparison: Zolpidem (Ambien) Treatment vs Mind-Body Bridging; Test type: Superiority or Other; p = 0.13, ANCOVA

ADVERSE EVENTS:
Arm/Group | Zolpidem (Ambien) Treatment | Mind-Body Bridging
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/41
Other Adverse Events (participants affected / at risk) | 0/31 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No